CLINICAL TRIAL: NCT07278492
Title: Nicotinamide Adenine Dinucleotide Augmentation to Prevent or Reverse the Progression of Alzheimer's Disease in People With Down Syndrome
Brief Title: NAD Augmentation to Prevent or Reverse Alzheimer's Disease in People With Down Syndrome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025p002197
Record Dates: First submitted 2025-11-24; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Down Syndrome (DS)
Keywords: Down Syndrome; NMN; safety
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo controlled multiple ascending dose trial of NMN in adults with DS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety and pharmacokinetic ascending dose intervention group (Experimental): MIB-626 tablets will be provided at dose strength of 500mg. Three doses will be studied in ascending order: 500 mg (one tablet) once daily; 1000 mg (two 500 mg tablets once daily) or 1000 mg (two 500 mg tablets) twice daily.
  Interventions: Drug: MIB-626
- Placebo tablets (Placebo Comparator): Matching placebo tablets (number and frequency of tablets will match the active intervention group at each of the three doses)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MIB-626 — MIB-626 tablets will be provided at dose strength of 500mg. Three doses will be studied in ascending order: 500 mg (one tablet) once daily; 1000 mg (two 500 mg tablets once daily) or 1000 mg (two 500 mg tablets) twice daily.
  Arms: Safety and pharmacokinetic ascending dose intervention group
Drug: Placebo — Matching placebo tablets (number and frequency of tablets will match the active intervention group at each of the three doses)
  Arms: Placebo tablets

SUMMARY:
The aim of the study is to determine the safety and tolerability of different increasing doses of MIB-626 (a microcrystalline form of β nicotinamide mononucleotide; NMN) given daily for 28 consecutive days to adults with Down syndrome (DS). The study will also explore how the drug moves through the body over time (pharmacokinetics or PK) and how the drug affects the body in different ways (pharmacodynamics or PD). The study participants will be monitored for adverse events and measurements to detect safety events will take place including laboratory tests of blood counts, chemistries and coagulation profile, and electrocardiogram (ECG). The trial will enroll a total of 24 adults with DS who are 18 years or older and are medically stable. People enrolled in the study will be randomly assigned to receive either the active intervention (MIB-626) tablets, or placebo tablets for 28 days. Study participants will be followed for an additional 28 days (total 56 days of follow-up). This study will also explore the effect of MIB-626 on different measures associated with aging and risk of Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Specific Aims / Objectives Primary Aim To determine the safety and tolerability of multiple ascending doses of MIB-626 administered daily for 28 consecutive days in adults with DS by structured monitoring of adverse events and the measurement of safety laboratory tests including blood counts and chemistries, coagulation profile, and ECG.

Secondary Aims

1. To study the PK of oral, multiple ascending doses of MIB-626 in adults with DS starting with the 500 mg daily dose and escalating the dose in ascending order to the maximum dose of 1000 mg twice daily or a maximal tolerated dose if that is lower than 1000 mg twice daily dose. PK parameters (Caverage 0-24 h, Cmax, Tmax, AUClast, AUC24hr, AUCinf, and T1/2) will be computed using nonparametric methods.
2. To characterize the pharmacodynamics (PD) of MIB-626 by analyzing the blood concentrations of NAD+ and plasma concentrations of NAD+ metabolites (nicotinamide, 1-methylnicotinamide, N-Methyl-2-pyridone-5-carboxamide [2-PY], N-Methyl-4-pyridone-3-carboxamide [4-PY], nicotinic acid, and nicotinuric acid). The concentrations in urine of NAD+ metabolites will also be measured. The investigators will determine whether oral MIB-626 increases the abundance of NAD+ in the brain, measured by ultra-high field 7T magnetic resonance spectroscopy (MRS).

Exploratory Aims This trial is neither long enough nor large enough to determine the effects of MIB-626 on Alzheimer's Disease (AD) imaging or plasma biomarkers, or neuropsychological outcomes. However, the investigators have included some clinically important exploratory outcomes: (1) blood pressure and lipids that were improved in earlier human studies with MIB-626, and which may independently affect morbidity, and mortality; (2) muscle performance and physical function because people with DS often experience physical limitations, and MIB-626 improves mitochondrial function and running distance in mice, and improves muscle fatigability in humans.

The trial will provide important information on the safety, PK, PD, and engagement of target mechanisms that is necessary for guiding the stepwise progression of this promising molecule towards larger efficacy trials.

Demonstration of Target Engagement

1. The concentrations of NAD and its metabolites in the PBMCs will be measured to determine the abundance of NAD in PBMCs.
2. The tissue concentrations of NAD in brain will be measured using the 7T MRS.

General Description of Study Design This is a Phase 1b, randomized, double-blind, placebo-controlled, multiple ascending dose study evaluating the safety, tolerability, PK and PD of MIB-626 in adults with DS. Approximately 24 participants aged 18 years and older will be enrolled. Participants will be assigned to up to three dose cohorts and will receive MIB-626 or placebo for 28 days. Safety, PK and PD assessments will be conducted throughout treatment and follow up periods.

Number of Centers: The study will be conducted at two trial sites: recruitment will take place at the Down Syndrome Program at the Mass General Hospital, and the study will be implemented at the Brigham and Women's Hospital.

Estimated Study Duration The study duration for each subject is anticipated to be up to about 12 weeks, which includes the screening, 4 weeks of intervention, and 28-day post-intervention follow-up visit after investigational product administration.

Subject Population: The participants (total n=24) will be adult men and women, 18 years or older, who have confirmed diagnosis of DS and are medically stable.

Doses, Dose Frequency, and Intervention Duration:

MIB-626 tablets will be provided at dose strength of 500 mg. Three dose levels will be studied: 500 mg (one tablet) once daily; 1000 mg (two 500 mg tablets once daily), or 1000 mg (two 500 mg tablets) twice daily.

Rationale for the Dosing Cohorts: Up to three dosing cohorts of 8 participants each will be studied successively in ascending order: 500 mg once daily, 1000 mg once daily, and 1000 mg twice daily. Within each dose cohort, 8 subjects will be randomized in a 3:1 ratio to receive either MIB-626 (n=6) or matching placebo (n=2) tablets daily for 28 consecutive days. The first cohort will receive either 500 mg MIB-626 or placebo once daily; the second cohort will receive 1000 mg MIB-626 or placebo once daily; and the third cohort will receive 1000 mg MIB-626 or placebo twice daily.

The selection of these dose levels was informed by the results of the previous single and multiple ascending dose studies in healthy adults without DS, as well as studies in middle-aged and older adults with metabolic disorders that demonstrated that MIB-626 doses from 500 mg once daily to 1000 mg twice daily are safe and well tolerated, and increase blood NAD+ levels in community dwelling healthy adults. Although in single ascending dose studies, a single 500 mg MIB-626 dose did not significantly raise blood NAD+ levels, other studies have shown that daily administration of MIB-626 doses as low as 250 mg daily consecutively for 4 or more weeks raised blood or PBMC NAD+ concentration above baseline; the increase in NAD+ levels at doses less than 500 mg daily was substantially smaller than that associated with 500 mg daily or higher doses.

Study Schema: The 8 eligible subjects at each dose cohort will be randomized to MIB-626 or placebo using concealed block randomization in a 3:1 ratio. The dose escalation will be sequential.

Subject Selection Study Subjects and Recruitment Methods The participants will be community-dwelling adults, 18 years or older, with a confirmed diagnosis of DS.

Participant Recruitment:. Participants will be recruited at the Down Syndrome Program of Massachusetts General Hospital and through outreach to the DS community. Recruitment efforts will include engagement with local clinics, community organizations and patient registries.

Participant Retention:

Participant retention will be supported through regular communication with participants and/or caregivers, and reminder visit notifications throughout the study. Study staff will remain available to address questions or concerns during participation. Furthermore, the participants will receive reminders of appointments, have pleasant clinic visits, limited waiting time and coordinated assessments.

Excluded Medications and Treatments:

The ingestion of the following is prohibited for the duration of the intervention period (through the last study visit):

* The following medications are prohibited: niacin or dietary supplements containing NMN or nicotinamide riboside; any products that contain niacin, nicotinic acid, nicotinamide in any form, other than natural foods
* Occasional use of acetaminophen and nonsteroidal anti-inflammatory drugs, such as ibuprofen, for fever or headache is permitted.
* The use of recreational drugs such as marijuana, cocaine, amphetamines, or other street drugs is not permitted for the duration of the study (through the last study visit).

The study is double-blind in that the study participants and the study staff involved in outcomes assessments will be unaware of the intervention assignment.

IRB Approval IRB must be constituted according to the applicable state and federal/local requirements of each participating region. The NIH or designee may require documentation noting all names and titles of members who make up the respective IRB. If any member of the IRB has direct participation in this study, written notification regarding his or her abstinence from voting must also be obtained. If the site is unwilling to provide names and titles of all members due to privacy and conflict of interest concerns, it should instead provide a Federal Wide Assurance Number or comparable number assigned by the Department of Health and Human Services.

The PI or designee will supply relevant documents for submission to the respective IRB for the protocol's review and approval. This protocol, the Investigator's Brochure, a copy of the informed consent form, and the subject recruitment materials and/or advertisements and other documents required by all applicable laws and regulations, must be submitted to the local IRB for approval. The IRB's written approval of the protocol and subject informed consent must be obtained and submitted to the NIH before commencement of the study (i.e., before shipment of the investigational drug or study specific screening activity). The IRB approval must refer to the study by exact protocol title, number, and version date; identify versions of other documents (e.g., informed consent form) reviewed; and state the approval date. The drug's manufacturer will ship drug/notify site once the PI has confirmed the adequacy of site regulatory documentation and, when applicable, the PI has received permission from competent authority to begin the trial. Until the site receives drug/notification no protocol activities, including screening may occur.

The site must adhere to all requirements stipulated by their respective IRB. This may include notification to the IRB regarding protocol amendments, updates to the informed consent form, recruitment materials intended for viewing by subjects, local safety reporting requirements, reports and updates regarding the ongoing review of the study at intervals specified by the respective IRB, and submission of the investigator's final status report to IRB..

Investigational Product and Materials Dosage Form, Manufacturing, Packaging, and Labeling: In this protocol, the investigational product refers to either the active product, MIB-626 or the placebo.

Investigational Product: The MIB-626 will be a GMP-grade microcrystalline solid NMN mixed with inert excipients (including microcrystalline cellulose) and compressed into tablets at a dose strength of 500 mg per tablet, enabling administration of the 500 mg once daily using one tablet taken once daily; 1000 mg using two 500-mg tablets once daily; and 2000 mg using two 500-mg tablets twice daily.

Metro International Biotech, LLC will provide the active drug and matching placebo tablets.

Storage The procedures for the shipment, receipt, storage, dispensing, and instructions on how to handle temperature excursions are provided in the Pharmacy Manual:

The investigational product will be kept in an appropriate, limited access, secure place within the Investigational Drug Service (IDS) at each of the participating trial sites. The investigational product will be stored under the conditions specified in the Pharmacy Manual and will remain in the original container until dispensed. A temperature log of the drug storage area will be maintained every day.

Dose and Regimen: The subjects in each dose cohort will be randomized to receive either the placebo or MIB-626 daily orally in a 3:1 ratio. The first cohort will receive the 500-mg dose daily and the dose escalation will be sequential and contingent upon meeting the pre-specified criteria for dose escalation.

Group 1 Dose regimen: 500 mg MIB-626 or placebo daily, Number of Tablets: One 500-mg MIB-626 or one placebo tablet, Frequency: Once daily Group 2 Dose Regimen: 1000 mg MIB-626 or placebo, Number of Tablets: Two 500-mg MIB-626 tablets or two placebo tablets, Frequency: Once daily Group 3 Dose Regimen: 2000 mg MIB-626 or placebo, Number of tablets: Two 500 mg MIB-626 tablets or two placebo tablets twice daily, Frequency:Twice daily The participants will be instructed to take the study medication at 12-hour intervals.

Overall Dose Escalation: Stopping Rules Dose escalation will be sequential and will proceed as long as no pre-defined stopping criteria are met. Enrollment to the next dose cohort will not commence until an evaluation by the DSMB of all available safety data on all subjects on that dose through day 28 of study supports escalation to the next cohort.

Dose escalation will be suspended pending additional evaluation or terminated if any of the following occur:

The DSMB recommends that dose escalation should be suspended or terminated.

1. Two or more subjects in a dose cohort experience a drug-related, treatment-emergent adverse event of Grade 2 or higher by National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Dose Limiting Toxicity [DLT] Dose).

The Maximal Tolerated Dose (MTD) for this study is defined as that dose at which no more than 1 out of 6 subjects in a cohort experiences a Dose Limiting Toxicity (DLT). If 2 or more subjects in a cohort experience a DLT or meet Dose Escalation Stopping Rules, MTD will have been exceeded and the next lower dose level will be regarded as the MTD.

The MPIs, after discussion with the DSMB, or the DSMB may recommend termination of dose escalation if they believe AEs and/or laboratory abnormalities indicate that higher doses would not be tolerated or would jeopardize the subjects' safety. Factors that must be considered for termination of dose-escalation include the frequency, severity, clinical significance, and possible causality and anticipated reversibility of all observed AEs and/or laboratory abnormalities for each specific dose group. If the Investigator and/or the DSMB believe based on the available data that greater than minimal toxicity could potentially be experienced by subjects at a higher dose level, dose escalation may be terminated. Criteria supportive of termination of dose escalation may range from an aggregate of more frequent mild and/or moderate AEs and/or laboratory abnormalities that suggest consistent effects on any one or multiple major organ system(s) to less frequent, but more severe effects on a specific organ system.

Overall Definition of Dose Limiting Toxicity (DLT)

1. Dose Limiting Toxicity is defined as the occurrence of any of the following in 2 or more drug-treated subjects within a given dose cohort: Any Grade 2 or higher hematological or non-hematological toxicity per NCI CTCAE version 5.0, or
2. Any absolute QTc > 480 msec, any increase in QTc > 30 msec from baseline < 480 msec or any evidence of new onset of serious cardiac arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of full trisomy for chromosome 21 or complete unbalanced translocation of chromosome 21, confirmed by karyotype analysis or clinical documentation.
2. 18 years or older
3. Participant has a caregiver/ informant who has direct contact with the participant >10 hours/ week and who can provide information about participant's health
4. Participant or Legal Authorized Representative is able to understand and willing to provide written informed consent and capable of completing study assessments.
5. In addition, female participants must Not be pregnant and not planning to become pregnant over the next 6 months.

Exclusion Criteria

1. Fasting morning UACR > 5,000 mg/ g creatinine
2. Other laboratory abnormalities:

   1. Has AST or ALT > 3 times the upper limit of normal
   2. eGFR < 30 mL/ min / 1.73 m2
   3. Hematocrit < 0.34 or > 0.50 L/L
3. A major adverse cardiovascular event in preceding 3 months
4. Participation in an investigational trial to evaluate pharmaceuticals or biologics within the past 3 months or 5 half-lives, whichever is shorter
5. Current alcohol or substance use disorder or dependence (DSM 5 criteria).
6. Major depressive disorder, bipolar disorder, schizophrenia, or current psychotic symptoms or behavioral problems that could interfere with study procedures.
7. An acute illness, including COVID-19, requiring hospitalization within the past 3 months or any acute illness, including COVID-19, within the past month.
8. Has a history of anaphylaxis from vitamin B3 derivatives
9. BMI > 42.5 kg/ m2
10. Non-ambulatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Baseline to 56 days after drug administration
  All treatment emergent adverse events
Treatment emergent serious adverse events | Baseline to 56 days after drug administration
  All treatment emergent serious adverse events

SECONDARY OUTCOMES:
Pharmacokinetics of NMN | Baseline to 56 days
  Circulating levels of NMN
Pharmacodynamics - steady state concentration of NAD+ in the brain | Baseline and Day 28
  steady stage concentration of NAD+ in the brain measured in situ using ultra-high field 7T magnetic resonance spectroscopy (MRS)
Pharmacodynamics - Blood NAD+ level | Baseline to Day 56
  Blood NAD+ level
Pharmacodynamics - Plasma concentrations of NAD+ metabolites | Pre-dose up to Day 28
  Plasma concentrations of major NAD+ metabolites (nicotinamide, 1-methylnicotinamide, N-Methyl-2-pyridone-5-carboxamide [2-PY])
Urine concentration of NAD+ | Day 1 and Day 28
  Concentrations of timed urine collections of the major NAD+ metabolites (2-PY, 4-PY, nicotinamide and 1-methylnicotinamide)
Blood pressure | Baseline to Day 56
  Change in blood pressure measured under standard conditions
Hemoglobin A1c (HbA1c) | Change from baseline to 28 days
  Change in HbAIc over the 28-day intervention period
Fasting glucose and insulin | Baseline to 28 days
  Change in fasting glucose and insulin over the 28-day intervention period
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Change from baseline to 28 days
  Change in HOMA-IR over the 28-day intervention period
Change in biomarkers of aging: Insulin Growth Factor 1 (IGF-1) | Baseline to 28 days
  Change in IGF-1
Change in biomarkers of aging: Triiodothyronine (T3) | Baseline to 28 days
  Change in T3
Change in biomarkers of aging: Tumor necrosis factor-alpha (TNF-alpha) | Baseline to 28 days
  Change in TNF-alpha
Change in biomarkers of aging: F2-isoprostanes (F2-IsoPs) | Baseline to 28 days
  Change in F2-IsoPs

OTHER OUTCOMES:
Muscle strength and endurance | Baseline to Day 28
  muscle strength measured by the number of repetitions to failure with leg press exercise
Physical Function | Baseline to Day 28
  Six-minute walk test, distance walked in 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shalender K Bhasin, MB, BS, Principal Investigator — Brigham and Women's Hosptial
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No